CLINICAL TRIAL: NCT07272863
Title: The Impact of BBTI on Cognition and Sleep Health in Older Adults With HIV
Brief Title: The Impact of Brief Behavioral Treatment for Insomnia Versus Brief Mindfulness Treatment on Cognition and Sleep Health in Adults (Age 50+) With HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other); National Institute on Aging (NIA) (NIH); NIH Office of AIDS Research (OAR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-07-8836; R01AG092240 (NIH)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Cognition; Aging; HIV
Keywords: insomnia; cognition; older adults; HIV; Alzheimer's Disease; brief behavioral treatment; randomized control trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Treatment for Insomnia (BBTI) (Experimental)
  Interventions: Behavioral: BBTI
- Brief Mindfulness Treatment (BMT) (Active Comparator)
  Interventions: Behavioral: BMT

INTERVENTIONS:
Behavioral: BBTI — 4-week intervention delivered via telephone (once a week for 30 minutes)
  Arms: Brief Behavioral Treatment for Insomnia (BBTI)
Behavioral: BMT — 4-week intervention delivered via telephone (once a week for 30 minutes)
  Arms: Brief Mindfulness Treatment (BMT)

SUMMARY:
The goal of this clinical trial is to examine the effects of a telephone-delivered Brief Behavioral Treatment Insomnia (BBTI) versus a Brief Mindfulness Treatment (BMT) on cognitive and sleep outcomes in older adults with HIV. The main questions it aims to answer are:

What are the effects of BBTI vs BMT on self-reported and observed sleep outcomes in older adults with HIV and insomnia up to 1-year post-intervention? What are the effects of BBTI vs BMT on self-reported and observed cognitive comes in older adults with HIV and insomnia up to 1-year post-intervention? What is the association between Alzheimer's Disease biomarkers and sleep and cognitive outcomes in older adults with HIV receiving BBTI vs BMT?

Participants will:

* Complete 4 weeks of telephone-delivered BBTI or BMT
* Attend baseline, post-intervention, and 1-year post in-person visits for sleep and cognitive assessments
* Have blood collected at all three time points

ELIGIBILITY:
Inclusion Criteria:

* must be age 50 or older
* have a DSM-5 diagnostic criteria for insomnia including sleep difficulty that occurs at least 3 times per week and has been a problem for at least 3 consecutive months (indicated on the Structured Clinical Interview for Sleep Disorders, SCISD) during telephone screening
* have a confirmed HIV diagnosis and a prescribed ART regimen for at least 12 months.

Exclusion Criteria:

* unable to speak English
* have a reported or documented (in medical records) diagnosis of AD or dementia
* have severe neurocognitive impairment (>7 errors on the Short Portable Mental Status Questionnaire, SPMSQ) during telephone screening
* have a history of a stroke
* currently undergoing radiation/chemotherapy
* reports a history of brain trauma with loss of consciousness greater than 30 minutes
* have a learning disability
* have a documented diagnosis of sleep apnea (in medical records)
* reports use of a continuous positive airway pressure machine
* have been identified as high risk for moderate to severe sleep apnea (Snoring, Tiredness, Observed sleep apnea, Pressure, BMI, Age, Neck circumference, and Gender, STOP BANG ≥ 5) during telephone screening
* have restless leg syndrome and/or have narcolepsy
* have a documented history of bipolar disorder or psychotic disorder
* not be receiving efavirenz as part of their current ART regimen

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | From enrollment until 1-year post-intervention
  Assesses insomnia severity symptoms with scores ranging from 0 - 28. Scores of 0-7 indicate no clinically significant insomnia; scores 8-14 indicate mild insomnia; scores 15-21 indicate moderate insomnia; scores 22-28 indicate severe insomnia
7-day Sleep Actigraphy | From enrollment until 1-year post-intervention
  Actigraphy will be conducted at (baseline, post-intervention. and 1-year post intervention) to obtain objective sleep data including total sleep time, falling asleep time, wake-up time, sleep latency, awakenings after sleep onset, and sleep efficiency.
Consensus Sleep Diaries | From enrollment until 1-year post-intervention
  The diaries will be completed twice a day (before going to bed at night, and then the following morning) in conjunction with the actigraphy measurement of their sleep to improve the quality of the actigraphy data.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | From enrollment until 1-year post-intervention
  Consists of 12 subtests measuring five domains: Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory. RBANS has four equivalent alternate test forms. Total scores range from 40 to 160, with higher scores indicating better cognitive function
Delis-Kaplan Executive Function System (D-KEFS) | From enrollment until 1-year post-intervention
  Three D-KEFS tests will be used for this study: Trail Making Test, Verbal Fluency Test, and Color-Word Interference Test.
Patient's Assessment of Own Functioning Inventory (PAOFI) | From enrollment until 1-year post-intervention
  Measures the effects of cognitive abilities on everyday activities. Scores are summed from each domain for a total score ranging from 0 to 50, with higher scores indicated worse perceived everyday functioning.
Pittsburgh Sleep Quality Index (PSQI) | From enrollment until 1-year post-intervention
  An 18-item questionnaire used to assess sleep quality. Scores from 7 components are summed for a global PSQI score range from 0-21, with higher scores (> 5) indicating poorer quality of sleep.

SECONDARY OUTCOMES:
Amyloid beta (Aβ42/40) | From enrollment until 1-year post-intervention
  Aβ42/40 ratio is a marker of amyloid plaque accumulation which is a hallmark of Alzheimer's Disease
P-tau | From enrollment until 1-year post-intervention
  Biomarker for identifying individuals at risk for Alzheimer's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shameka L Cody, PhD, AGNP-C, PMHNP-BC, FAAN, Principal Investigator — The University of Alabama Capstone College of Nursing
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Alabama, Tuscaloosa, Alabama

IPD SHARING:
Plan to Share IPD: No
The data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to use the data only for research purposes and not to identify any individual person; (2) a commitment to secure the data using appropriate computer technology; and (3) a commitment to destroy or return the data after analyses are completed. Although it is assumed that most users will want either a SAS or SPSS file, we have the ability to translate data sets into several other formats and will provide one of these if requested by a user

REFERENCES:
- [Background] Cody SL, Kusko DA, Gonzalez CE, Owens MA, Hobson JM, Gilstrap SR, Thomas SJ, Goodin BR. Improving Sleep in People with HIV and Chronic Pain: A Pilot Study of Brief Behavioral Treatment for Insomnia. Behav Sleep Med. 2024 Nov-Dec;22(6):949-959. doi: 10.1080/15402002.2024.2396820. Epub 2024 Sep 8. PMID 39244666